CLINICAL TRIAL: NCT04024319
Title: Ultrasound-guided Genicular Nerve Block an Analgesic Alternative to LIA for Total Knee Arthroplasty: Case-control Series
Brief Title: Ultrasound-guided Genicular Nerve Block for Total Knee Arthroplasty (GenTKR)
Acronym: GenTKR
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Xavier Sala-Blanch, Principal Investigator, Hospital Clinic of Barcelona
Other Study IDs: HCB/2018/0463
Record Dates: First submitted 2019-07-15; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Pain, Postoperative; Knee Pain Chronic
Keywords: Total Knee Replacement; Genicular nerves block; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Genicular Nerve Block: GNB will be performed on this group of patients undergoing TKR. The patient will be positioned in the supine position, with the extremity to operate slightly in external rotation. The anesthesiologist will be located ipsilateral to the knee to intervene; asepsis will be performed with 70% chlorhexidine, sterile gloves will be used and the ultrasound probe will be protected with a sterile cover. The ultrasound transducer will be placed in a long axis of the knee in the corresponding area to block according to anatomical repairs. 4 ml of 0,2% ropivacaine was administered in each GN.
  Interventions: Procedure: Genicular Nerve Block
- Local Infiltration Analgesia: Retrospectively, the data of the patients belonging to the control group (LIA) were collected through the electronic file in the SAPP program of the internal network of the Barcelona Clinic Hospital in chronological order until completing 35 cases. To include them in the control group, the patients had to meet the same criteria as those belonging to the intervention group (GNB), therefore, the surgery should have been performed under spinal anesthesia and subsequently followed with an oral analgesia schedule meeting criteria of fast track hospitalization. The same data were obtained as in the GNBG, demographic data (age, sex, weight, height, hematocrit, hemoglobin, ASA), duration of the surgery and ischemia time, PACU VAS, AM VAS, PM VAS and finally some data of the post-operative period (hematocrit, hemoglobin, transfusion, hospital stay)

INTERVENTIONS:
Procedure: Genicular Nerve Block — 4 ml of local anesthetic were administered in 5 genicular nerves. A total volume of 20 ml were administered in GNB group.
  Groups: Genicular Nerve Block

SUMMARY:
Knee Osteoarthritis affects one third of the population over 65 years old. Total knee arthroplasty (TKA) has become one of the most frequent surgical procedures in the world. During the last years it went from being a long hospital stay surgery to a fast track procedure. Currently models employ high volume local infiltration techniques (LIA). The genicular nerve block (GNB) appears as alternative in this patients.

The objective of this study is to evaluate the analgesic results of genicular nerve block after TKA in a small cohort of patients.

35 patients scheduled for TKA underwent to GNB were included. Pain measurement.

DETAILED DESCRIPTION:
An observational study of a series of 35 cases will be carried out based on the casuistry of TKR surgery of the investigator's center. The performance of analgesic blockade called GNB in adult patients, ASA physical status I-III, which will undergo TKR, will be part of the multimodal analgesia strategy.

After compliance with the inclusion criteria, with the acceptance and signature of the informed consent by the participating patients, the following procedure will be followed:

1. Patients will be routinely assessed by an anesthesiologist of the service, later they will enter the operating room, where the vital signs will be monitored and the usual anesthetic technique will be used for TKR, that is, spinal anesthesia.
2. To perform the blocks a 90 mm needle was used, with a 30mm extension connected to a 20ml syringe with a mixture of 20ml of 0.2% ropivacaine + 200 micrograms of adrenaline. The needle will be advanced with an out-of-plane technique and 4 ml of the described solution will be placed in each of the 5 nerves to be blocked: Superomedial genicular nerve (SMGN), Superolateral genicular nerve (SLGN), Inferomedial genicular nerve (IMGN), Inferolateral genicular nerve (ILGN) and Recurrent tibial genicular nerve (RTGN) .
3. The pain assessment will be carried out during the night after the intervention (approximately 12 hours) and the next morning (approximately 24 hours). The pain will be objectified by (VAS) (0-10) by a nurse, blind to the analgesic treatment. The use of rescue opioids will be indicated in case of VAS ≥ 3, data that will also be analyzed. In the room, the pharmacological treatment established as an institutional protocol will continue. It should be noted that these data as well as demographic data, intraoperative times, and relevant post-operative data (hematocrit, complication) were obtained from the clinical records of the electronic file of the program used in the internal network of the Barcelona Clinic Hospital
4. Researchers will record those variables aimed at evaluating the intensity of acute postoperative pain 24 hours after TKR (Pain score ≥ 4 in any time).

These results will be included, anonymously, in an Excel database made for this purpose for further analysis. The variables will be recorded in a single intervention

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing TKR
* Acceptance to participate
* ASA physical status II-III
* Age > 18 years

Exclusion Criteria:

* Refusal to participate in the study
* Allergy to local anesthetics
* History of substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing TKR in Hospital Clinic
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Maximum Pain score in first day after surgery | 48 hours
  Post operative pain scores will be recorded with a NRS(numerical rating scala) from 0 to 10 ( 0=no pain, 10= pain as bad as can be) worst score at 12 hrs, 24 hrs and 48 hrs period will be scored.

CONTACTS AND LOCATIONS:
Overall Officials: xavier sala-blanch, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pietrantoni P, Cunat T, Nuevo-Gayoso M, Martin N, Tio M, Basora M, Sastre S, Sala-Blanch X. Ultrasound-guided genicular nerves block: an analgesic alternative to local infiltration analgesia for total knee arthroplasty: A noninferiority, matched cohort study. Eur J Anaesthesiol. 2021 Aug 1;38(Suppl 2):S130-S137. doi: 10.1097/EJA.0000000000001546. PMID 34038916